CLINICAL TRIAL: NCT04825366
Title: Restoration of Hypoglycemia Awareness With Home-based High Intensity Interval Training in Adults With Type 1 Diabetes and Impaired Awareness of Hypoglycemia
Brief Title: Restoration of Hypoglycemia Awareness With Home-based High Intensity Interval Training
Acronym: FEEL-HIIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Full professor, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-1117
Record Dates: First submitted 2021-03-28; First posted 2021-04-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Type 1 Diabetes; Hypoglycemia Unawareness
Keywords: Type 1 diabetes; Hypoglycemia unawareness; Education; Avoidance of hypoglycemia; High intensity interval training
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Continuous Glucose Monitoring; Health; Heart Rate Determination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard educational program (Active Comparator): Participants will be closely followed by a team of diabetes specialists. Participants will attend two education sessions to discuss the following topics: avoidance of hypoglycemia, causes of hypoglycemia, treatment (e.g. glucagon) of hypoglycemia, how to better recognize hypoglycemia symptoms, understand how to use a continuous glucose monitor (CGM) and understand CGM reports to adjust insulin doses.
  Interventions: Device: Continuous glucose monitoring device; Other: Gold method; Other: Clarke questionnaire; Other: Edinburgh Hypoglycemia Symptom Scale; Other: BAPAD questionnaire; Other: Hypoglycemia Fear Survey II; Other: Physical activity questionnaire; Other: Well-being; Other: Treatment satisfaction; Other: Hypoglycemia diary; Device: Piezo RxD
- Standard educational program combined with high intensity interval training (Active Comparator): Participants will be closely followed by a team of diabetes specialists. Participants will attend two education sessions to discuss the following topics: avoidance of hypoglycemia, causes of hypoglycemia, treatment (e.g. glucagon) of hypoglycemia, how to better recognize hypoglycemia symptoms, understand how to use a continuous glucose monitor (CGM) and understand CGM reports to adjust insulin doses.
  Each study participant will be asked to train 3 times per week following the home-based program that will be provided to them. Participants will be asked to perform at least 2 training sessions per week with the exercise specialist on a virtual platform. The training session will consist of a 3 to 5-minute low-intensity warm-up followed by 6 to 12 1-minute bouts of high-intensity exercise interspersed with 1-minute bouts of low-intensity exercise. Each session will end with a 3-minutes cool-down period.
  Interventions: Device: Continuous glucose monitoring device; Other: Gold method; Other: Clarke questionnaire; Other: Edinburgh Hypoglycemia Symptom Scale; Other: BAPAD questionnaire; Other: Hypoglycemia Fear Survey II; Other: Physical activity questionnaire; Other: Well-being; Other: Treatment satisfaction; Other: Hypoglycemia diary; Device: Piezo RxD; Device: Heart rate monitor; Other: Exercise diary

INTERVENTIONS:
Device: Continuous glucose monitoring device — Participants will have to wear their continuous glucose monitoring device throughout the study.
Other: Gold method — The Gold method will be used to assess impaired awareness of hypoglycemia
Other: Clarke questionnaire — The Clarke questionnaire will be used to assess impaired awarness of hypoglycemia
Other: Edinburgh Hypoglycemia Symptom Scale — The Edinburgh Hypoglycemia Symptom Scale will be used to assess symptoms of hypoglycemia
Other: BAPAD questionnaire — The BArriers to Physical Activity in type 1 Diabetes (BAPAD) questionnaire will be used to assess barriers of physical activity
Other: Hypoglycemia Fear Survey II — The Hypoglycemia Fear Survey II will be used to assess fear of hypoglycemia
Other: Physical activity questionnaire — The International Physical Activity Questionnaire will be used to assess physical activity practice
Other: Well-being — The WHO-5 well-being index will be used to assess well-being.
Other: Treatment satisfaction — The Diabetes Treatment Satisfaction Questionnaire will be used to assess treatment satisfaction.
Other: Hypoglycemia diary — Participants will be asked to record in a diary treatments for hypoglycemic events
Device: Piezo RxD — Participants will be asked to wear a pedometer throughout the study
Device: Heart rate monitor — During training sessions, participants will be asked to wear a heart rate monitor
  Arms: Standard educational program combined with high intensity interval training
Other: Exercise diary — Before each training session, participants will be asked to note in a diary their glucose levels, if they have taken a snack or not and if insulin was administered. After each training session, participants will be asked to note that same information. In addition, they will be asked to note their bedtime blood glucose, if they have taken a bedtime snack and if adjustment to insulin doses was made.
  Arms: Standard educational program combined with high intensity interval training

SUMMARY:
The objective of this study is to investigate if the addition of a 12-week program of home-based high intensity interval training to a standard educational program aiming at preventing hypoglycemia episodes will restore hypoglycemia awareness in people living with type 1 diabetes and impaired awareness of hypoglycemia to a further extent than a standard educational program alone.

Participants will be randomized for 12 weeks to the standard educational program with or without high intensity interval training. The Gold method will be used to identify people with impaired awareness of hypoglycemia.

The educational program will consist of two education sessions on avoidance of hypoglycemia, causes of hypoglycemia, treatment (e.g. glucagon) of hypoglycemia, how to better recognize hypoglycemia symptoms, understand how to use a CGM/Flash-GM and understand CGM/Flash-GM reports to adjust insulin doses.

Participants randomized to the training program will be asked to train three times per week for 12 weeks following the home-based program that will be provided to them. Participants will be asked to perform at least 2 training sessions per week (ideally all 3 sessions) with the exercise specialist on a virtual platform.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged between 18 and 65 years old.
2. Clinical diagnosis of type 1 diabetes for at least five years.
3. Treatment with multiple daily insulin injections or insulin pump therapy and using insulin analogs (rapid, ultra-rapid or basal). The type of insulin should be stable for at least 1 month. Participants not using an insulin analog will be offered the opportunity to switch to an insulin analog and this will be done at least 1 month before inclusion.
4. Impaired awareness of hypoglycemia (Gold score ≥ 4).
5. HbA1c ≤ 10%
6. Using a continuous glucose monitor or being willing to start using one for the study
7. Having an electronic device supporting the Polar Beat application (heart rate monitor).

Exclusion Criteria:

1. Clinically significant microvascular complications: nephropathy (estimated glomerular filtration rate below 40 ml/min), neuropathy (especially advanced peripheral neuropathy with significantly lower limb reduced proprioceptive perception) or severe proliferative retinopathy as reported by the patient and/or judged by the investigator.
2. High risk foot problem (e.g., previous amputation, history of foot wound, known severe neuropathy or peripheral arterial disease)
3. Recent (< 3 months) acute macrovascular event e.g., acute coronary syndrome or cardiac surgery or history of significant heart disease.
4. Known significant cardiac rhythm abnormality based on investigator judgment.
5. Abnormal blood panel and/or anemia (Hb < 100g/L).
6. Ongoing pregnancy or breastfeeding.
7. Severe hypoglycemic episode or diabetic ketoacidosis within 1 month of screening.
8. Uncontrolled hypertension (blood pressure >160/100 mm Hg).
9. Uncontrolled angina.
10. Treatment with oral steroids within the last 3 months.
11. History of significant lung disease that would limit exercise.
12. Seizure within the last 3 months.
13. Participation in high-intensity interval training (or equivalent) in the past 6 months.
14. Physical ability preventing the completion of the 12-week training program (e.g., orthopedic limitation).
15. Inability to give consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Change in the Gold score | 12 weeks
  The Gold method is used to assess impaired awareness of hypoglycemia. The scale is from 1 to 7. A score of 4 or more indicates impaired awareness of hypoglycemia

SECONDARY OUTCOMES:
Change in the Clarke score | 12 weeks
  The Clarke questionnaire is used to assess impaired awareness of hypoglycemia. The scale is from 0 to 7. A score of 4 or more indicates impaired awareness of hypoglycemia
Change in the score of the Edinburgh Hypoglycemia Symptom Scale | 12 weeks
  Symptoms of hypoglycemia
Change in the score of the BAPAD questionnaire | 12 weeks
  Barriers to physical activity. The score can be between 12 and 84. A higher score means more barriers to physical activity.
Change in the score of the Hypoglycemia Fear Survey II | 12 weeks
  Fear of hypoglycemia. The score can be between 0 and 132. A higher score means higher level of fear of hypoglycemia.
Change in physical activity practice | 12 weeks
  Score of the International Physical Activity Questionnaire
Change in well-being | 12 weeks
  Score of the WHO-5 well-being index. The score can be between 0 and 5. Higher scores means better well-being.
Change in treatment satisfaction | 12 weeks
  Score of the Diabetes Treatment Satisfaction questionnaire. The score can be between 0 and 36. Higher score means better satisfaction.
Percentage of participants who no longer have impaired awareness of hypoglycemia | 12 weeks
Percentage of time of glucose levels spent < 4.0 mmol/L | 12 weeks
  Based on continous glucose monitor data
Percentage of time of glucose levels spent < 3.0 mmol/L | 12 weeks
  Based on continous glucose monitor data
Percentage of time of glucose levels spent between 3.9-10.0 mmol/L | 12 weeks
  Based on continous glucose monitor data
Percentage of time of glucose levels spent > 10.0 mmol/L | 12 weeks
  Based on continous glucose monitor data
Standard deviation of glucose levels | 12 weeks
  Based on continous glucose monitor data
Coefficient of variation of glucose levels | 12 weeks
  Based on continous glucose monitor data
Number of hypoglycemic events | 12 weeks
  Glucose levels < 4 mmol/L or < 3 mmol/L
Number of treated hypoglycemic events | 12 weeks
  Number of time that carbohydrates were taken to treat a hypoglycemia event
Number of severe hypoglycemia | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada